CLINICAL TRIAL: NCT06746142
Title: Free Breathing Versus Deep Inspiration Breath Hold Technique in Adjuvant Radiotherapy for Left Sided Breast Cancer: A Dosimetric Comparison of Target Volumes, Heart and Left Lung
Brief Title: Dosimetric Comparison of Target Volume, Heart and Left Lung in Post Mastectomy Radiotherapy (RT) of Left Sided Breast Cancer by Free Breathing (FB) Versus Deep Inspiration Breath Hold (DIBH) Technique
Acronym: FB DIBH RT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nishat Tasnim (Other)
Collaborators: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Sponsor-Investigator, Nishat Tasnim, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Organization: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5104
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma Breast; Radiation Therapy for Primary Breast Cancer; Radiation Tolerance; Radiation Induced Cardiac Damage; Radiation Induced Lung Injury (RILI); Radiotherapy; Adverse Effect; Radiotherapy, Adjuvant
Keywords: Deep Inspiration Breath Hold Technique; Post mastectomy radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A: FB RT arm (Experimental): Participants will be treated with 40.05 Gy radiation, at 2.67 Gy daily single fraction, 5 days a week, for 3 weeks by IMRT in free breathing technique.
  Interventions: Radiation: Free breathing radiotherapy
- Arm B: DIBH RT arm (Experimental): Participants will be treated with 40.05 Gy radiation, at 2.67 Gy daily single fraction, 5 days a week, for 3 weeks by IMRT in DIBH technique.
  Interventions: Radiation: Deep inspiration breath hold radiotherapy

INTERVENTIONS:
Radiation: Deep inspiration breath hold radiotherapy — Participants will be trained for 2-3 days for obtaining the desired breathing cycle by trained technologists. No extra equipment will be needed. At first, they will be assured and asked to relax. Then instructed to breath in and out twice followed by a slow, deep breath in to a comfortable higher level than normal and to hold it for at least 20 seconds then again breath normally. Once they are ready with expected breath holding, simulation will be done. Treatment will also be given in this breath holding position.
  Arms: Arm B: DIBH RT arm
Radiation: Free breathing radiotherapy — Patient will be advised for free breathing during simulation and treatment.
  Arms: Arm A: FB RT arm

SUMMARY:
Breast cancer is a leading cancer among Bangladeshi female. For breast cancer, there are different available treatment options according to the stage of disease. One of the important ones is radiotherapy (RT). Various side effects can occur during and after RT. Among the late side effects, numerous cardiac and pulmonary problems are significant specially in case of left sided breast cancer. In such cases, patients are being cured from cancer but the treatment itself endangering patients' general health and wellbeing by increasing risk of future life threatening cardiac and pulmonary diseases. Studies from around the world have shown that, during RT of left sided breast cancer, holding the breath for certain time after deep inspiration can reduce the radiation doses to heart and left lung without compromising doses to the chest wall. As a result, they can avoid the extra risk of treatment related late toxicities. This study will look at the utility and efficacy of Deep Inspiration Breath Hold (DIBH) RT over free breathing (FB) RT in reducing the heart and left lung doses without compromising the dose to the target volumes in left sided post mastectomy breast cancer patient, which is the main objective of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven left sided invasive breast cancer patients who underwent modified radical mastectomy.
2. Post mastectomy patients for whom radiotherapy including supraclavicular irradiation is indicated.
3. Patients having ECOG performance status up to 1.

Exclusion Criteria:

1. Left sided breast cancer patient underwent BCS.
2. Patient received any chemotherapy other than Doxorubicin, Cyclophosphamide and taxane (Paclitaxel/ Docetaxel) in any settings (neoadjuvant or adjuvant).
3. Patients who have comorbidities that would hinder DIBH (extreme obesity, mental disorder, hypoacusis etc.).
4. Known case of patients with respiratory diseases.
5. Known case of patients with ischemic heart diseases.
6. Patients with previous history of radiotherapy to chest.
7. Male breast cancer patients.
8. Bilateral breast cancer patients.
9. Pregnant or lactating women.
10. Age ˂ 18 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Radiation dose to target volume, left lung and heart | Immediately after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Most. Rokaya Sultana, MBBS, MD, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (4):
- Bangladesh (4):
  - Bangabandhu Sheikh Mujib Medical University, Dhaka
  - Combined Military Hospital, Dhaka, Dhaka
  - Delta Hospital Limited, Dhaka, Dhaka
  - Lab Aid Cancer Hospital, Dhaka, Dhaka

DOCUMENTS (1):
  • Study Protocol (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06746142/Prot_000.pdf